CLINICAL TRIAL: NCT00892671
Title: Airway Management and Vascular Access Simulation
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Thomas R. Vetter, PI, UAB Department of Anesthesiology
Other Study IDs: E080829003
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2010-08

CONDITIONS: Airway Management; Vascular Access
Keywords: Perceived effectiveness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- medical students
  Interventions: Other: Simulation

INTERVENTIONS:
Other: Simulation — simulation of airway management and vascular access

SUMMARY:
This project involves a pre- and post- airway management and vascular access simulation survey. The purpose of the study is to assess the perceived effectiveness of the simulation course on the performance of medical students enrolling in the Anesthesiology rotation during their third and fourth year of medical education.

ELIGIBILITY:
Inclusion Criteria:

* medical student enrolled in the Department of Anesthesiology rotation

Exclusion Criteria:

* anyone not enrolled in the rotation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: third and fourth year medical studens enrolling in the UAB Department of Anesthesiology rotation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
perceived effectiveness | pre- and post- simulation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Vetter, MD, MPH, Principal Investigator — University of Alabama at Birmingham Department of Anesthesiology
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States